CLINICAL TRIAL: NCT05951205
Title: A Phase 3 Study to Evaluate Efficacy and Safety of a Single Dose of Exa-cel in Subjects With Severe Sickle Cell Disease, βS/βC Genotype
Brief Title: Evaluation of Efficacy and Safety of a Single Dose of Exa-cel in Participants With Severe Sickle Cell Disease, βS/βC Genotype
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX21-CTX001-171; 2023-503247-34-00 (Other: EU CT number); 2021-006375-41 (EudraCT Number)
Record Dates: First submitted 2023-06-23; First posted 2023-07-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — exagamglogene autotemcel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Exa-cel (Experimental): Participants will receive a single infusion of exa-cel (autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the erythroid lineage-specific enhancer of the BCL11A gene) through a central venous catheter.
  Interventions: Biological: Exa-cel

INTERVENTIONS:
Biological: Exa-cel — Administered by intravenous (IV) infusion following myeloablative conditioning with busulfan.
  Other Names: Exagamglogene autotemcel; CTX001

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of CTX001 (exa-cel) in adolescent and adult participants with severe sickle cell disease (SCD), βS/βC genotype (HbSC).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with documented βS/βC (HbSC) genotype
* Participants must be eligible for autologous stem cell transplant as per investigator's judgment

Key Exclusion Criteria:

* A willing and healthy 10/10 human leukocyte antigen (HLA)-matched related donor is available per investigator's judgement
* Participants with prior hematopoietic stem cell transplant (HSCT)
* Treatment with regular RBC transfusions that, in the opinion of the investigator, cannot be interrupted after engraftment.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2027-07-31 (Estimated); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with an Average Fetal Hemoglobin (HbF) Greater Than or Equal To (>=) 20 percent (%) on or After 6 Months | From 60 Days after Last Red Blood Cell (RBC) transfusion up to 24 Months after exa-cel infusion

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent up to 24 Months After exa-cel Infusion
Proportion of Participants With Neutrophil Engraftment (First day of 3 Consecutive Measurements of Absolute Neutrophil Count (ANC) >=500 per Microliter [mcgL] on 3 Different Days) | Within 42 Days After exa-cel Infusion
Time to Neutrophil Engraftment | Up to 24 months After exa-cel Infusion
Time to Platelet Engraftment | Up to 24 months After exa-cel Infusion
Incidence of Transplant-Related Mortality (TRM) | Up to 100 Days After exa-cel Infusion
Incidence of Transplant-Related Mortality (TRM) | Within 12 Months After exa-cel Infusion
Incidence of All-cause Mortality | From Signing of Informed Consent up to 24 Months After exa-cel Infusion
Proportion of Participants With No Severe Vaso-Occlusive Crises (VOCs) for At least 12 Months (VF12) | From 60 Days after Last RBC transfusion up to 24 Months After exa-cel Infusion
Proportion of Participants Free from Inpatient Hospitalization For Severe VOCs Sustained for At least 12 Months (HF12) | From 60 Days after Last RBC transfusion up to 24 Months After exa-cel Infusion
Relative Reduction in Annualized Rate of Severe VOCs | From Baseline up to 24 Months After exa-cel Infusion
Duration of Severe VOC Free in Participants who Have Achieved VF12 | From 60 Days after Last RBC transfusion up to 24 Months After exa-cel Infusion
Relative Reduction in Rate of Inpatient Hospitalizations for Severe VOCs | From Baseline up to 24 Months After exa-cel Infusion
Relative Reduction in Annualized Duration of Hospitalization for Severe VOCs | From Baseline up to 24 Months After exa-cel Infusion
Proportion of Participants With Sustained HbF >= 20 % for At least 3, 6, or 12 months | From 60 Days after Last RBC transfusion up to 24 Months After exa-cel Infusion
Relative Reduction in Annualized Volume of RBC Transfusions | From Baseline Up To 24 Months After exa-cel Infusion
HbF Concentration Over Time | Up To 24 Months After exa-cel Infusion
Total Hemoglobin (Hb) Concentration Over Time | Up To 24 Months After exa-cel Infusion
Change In Reticulocyte Count Over Time | From Baseline Up To 24 Months After exa-cel Infusion
Change in Indirect Bilirubin Over Time | From Baseline Up To 24 Months After exa-cel Infusion
Change in Haptoglobin Over Time | From Baseline Up To 24 Months After exa-cel Infusion
Change in Lactate dehydrogenase (LDH) Over Time | From Baseline Up To 24 Months After exa-cel Infusion
Time to First Detectable Haptoglobin | Up to 24 Months After exa-cel Infusion
Time to First Normalized LDH | Up to 24 Months After exa-cel Infusion
Proportion of Alleles With Intended Genetic Modification Present in Peripheral Blood Over Time | Up To 24 Months After exa-cel Infusion
Proportion of Alleles With Intended Genetic Modification Present in CD34+ Cells of the Bone Marrow Over Time | Up To 24 Months After exa-cel Infusion
Change in Pain Scale (11-point numerical rating scale (NRS)) Assessment Over Time In Adults (>=18 Years) | From Baseline Up To 24 Months After exa-cel Infusion
Change in Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Over Time In Adults (>=18 Years) | From Baseline Up To 24 Months After exa-cel Infusion
Change in Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) | From Baseline Up To 24 Months After exa-cel Infusion
Change in Pain Scale (11-point NRS) Assessment Over Time In Adolescents (12 to <18 years of age) | From Baseline Up To 24 Months After exa-cel Infusion
Change in Pediatric Quality of Life Inventory (PedsQL; self-report and parent proxy versions) Generic Core In Adolescents (12 to <18 years of age) | From Baseline Up To 24 Months After exa-cel Infusion
Change in PedsQL SCD module (self-report and parent proxy versions) In Adolescents (12 to <18 years of age) | From Baseline Up To 24 Months After exa-cel Infusion

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing